CLINICAL TRIAL: NCT04981600
Title: LaseRF Trial: Radiofrequency Ablation vs. Laser Hemorrhoidoplasty Procedure for Grade II-III Hemorrhoidal Disease: Prospective Randomised Controlled Trial
Brief Title: LaseRF Trial: Radiofrequency Ablation vs. Laser Hemorrhoidoplasty for Hemorrhoidal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Collaborators: Istanbul Medipol University Hospital (Other); Gama Medical Ltd. (Unknown)
Responsible Party: Principal Investigator, Hanife Seyda Ulgur, Assistant Doctor, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/183
Record Dates: First submitted 2021-07-04; First posted 2021-07-29 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Hemorrhoids
Keywords: Radiofrequency ablation; Laser hemorrhoidoplasty; Pain; Recurrence
MeSH Terms: conditions — Hemorrhoids; Pain; Recurrence | interventions — Radiofrequency Ablation; Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Group (Active Comparator): Grade II-III hemorrhoids present a special challenge to surgeons since aggressive surgery exposes the patient to several per- and postoperative complications. Therefore new techniques have been developed and one of the most popular contemporary technique is laser hemorrhoidectomy. By this technique a laser probe is inserted above the dentate line and advanced to the apex of the cushion and several shots are delivered while pulling out the probe gradually. The idea is to compromise the vascular flow of corpus cavernosum recti, hence shrinking the hemorrhoidal cushion.
  Interventions: Device: Laser
- RF (Radiofrequency) Group (Active Comparator): Another recent and similar method is radiofrequency coagulation which depends on transmitting radiofrequency waves to tissue. This transmission results in conversion of radiofrequency waves into heat and causes coagulation necrosis in corpus cavernosum recti. The necrosis leads to fibrosis of the surrounding vessels and consequently cushion shrinkage is achieved.
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Radiofrequency ablation — Patients in the RF group will be first examined under anesthesia at the beginning of the procedure in lithotomy position. Approximately 3-6 ml of 20 mg/ml Lidocaine (Jetokaine, Adeka İlaç Sanayi, Samsun) solution will be injected between the cushion and the internal anal sphincter to minimize heat conduction to the surrounding tissues during the procedure. The HPR45i probe (F Care Systems, Antwerpen, Belgium) connected to the Rafaelo ® EVRF machine (F Care Systems, Antwerpen, Belgium) will be placed inside the cushion and 25 watts of RF energy will be transmitted. Care will be taken by not exceeding the dentate line caudally. The recommended Joule value for each operation is 1200-3000 J. Then cold is applied on the cushion, reducing the temperature of the tissue and preventing damage to the surrounding tissues. The same procedure will be performed for other pathologic cushions as well.
  Arms: RF (Radiofrequency) Group
Device: Laser — The same preoperative preparations will be done for the laser group as well. The NeoV 1470 (neoLaser, Israel) device will be used in this group. Following routine placement of the patient in lithotomy position and determining the cushion to be treated, a 12 W laser beam with a wavelength of 1470nm will be inserted into the cushion above the dentate line and advanced to the apex and approximately 3 laser shots are delivered throughout the course caudally, the number of which can be altered according to the size targeted cushion. Finally the procedure will be completed after gentle cold application.
  An enema will be given to the patients in both study groups in the morning of the operation and patients will be discharged with analgesics on the same day.
  Arms: Laser Group

SUMMARY:
Hemorrhoids, which can be defined as "vascular cushions" located at the anorectal junction, constitute an important part of the physiological continence mechanism. However, under various pathological conditions, they can expand below the dentate line and consequently are defined as hemorrhoidal disease, which is characterized by various symptoms such as bleeding, pain and itching. An ideal treatment should be effective in the long term, require less intervention to the surrounding structures, have low morbidity rates and cause minimal postoperative pain, which significantly affects the quality of life of a patient following surgery. he aim of this study is to compare the two contemporary minimally invasive methods.

DETAILED DESCRIPTION:
Hemorrhoids, which can be defined as "vascular cushions" located at the anorectal junction, constitute an important part of the physiological continence mechanism. However, under various pathological conditions, they can expand below the dentate line and consequently are defined as hemorrhoidal disease, which is characterized by various symptoms such as bleeding, pain and itching. The indication of treatment depends primarily on the individual burden of the disease rather than its stage. An ideal treatment should be effective in the long term, require less intervention to the surrounding structures, have low morbidity rates and cause minimal postoperative pain, which significantly affects the quality of life of a patient following surgery. Although conventional resection based techniques have less recurrence rates, they tend to have a greater chance of leading to various postoperative complications such as significant postoperative pain, urinary retention, bleeding, abscess formation, anal stenosis, anal fissure and fecal incontinence, deeming non-resection based less invasive techniques more favorable in terms of postoperative morbidity. The main mechanism of non-resection based techniques is creating an inflammatory stimulus inside the prolapsed hemorrhoidal tissue which ultimately causes fibrosis and relocation of the tissue above the dentate line. There are several randomized controlled trials which compared the laser procedure especially with resection based methods in this regard. However, to our knowledge, which is based on a thorough search in the Pubmed and Google Scholar, no randomized clinical trial has been made comparing the radiofrequency ablation method with the laser ablation technique .

The aim of this study is to compare the two contemporary minimally invasive methods in terms of postoperative complications, recovery process and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients who applied to the general surgery outpatient clinic due to stage 2 or 3 hemorrhoidal disease, unresponsive to medical treatment
* Patients who have not undergone any previous surgery due to hemorrhoidal disease
* Patients with written informed voluntary consent forms

Exclusion Criteria:

* Concomitant anorectal disease
* History of anticoagulant use
* Fecal incontinence complaint
* History of active steroid/immunosuppressive use for any reason
* Pregnancy
* Inflammatory Bowel Disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Rate of Healing | 4 month
  Hemorrhoid downgrading of at least 1 grade
Change in Visual analog score (VAS) at 4 weeks | 1st week and 4th week
  Patients are simply asked to score their pain from 1 to 10, which is typically called visual analog scale in the literature, with higher scores representing more severe pain.

SECONDARY OUTCOMES:
Quality of Life for HSS (Hemorrhoid Severity Score) | 1st week and 4th week
  Hemorrhoid Severity Score (HSS) is the total score obtained by the sum of the numerical grades of pruritis, pain, prolapse, bleeding and soiling. All the five components in this classification system are graded into four grades ranging from 0 to 3.
Operation Time | Operation 1 Day
  Specified in hours
Hospitalization Time | Discharge day after the surgery up to 3 days
  Specified in days
Number of admissions | 4 months after the procedure
  Outpatient follow up per routine or due to several complications such as pain, mucosal discharge, itching etc.
Rate of complications | 1st week, 4th week and 4th month
  Such as bleeding, infection and hematoma

CONTACTS AND LOCATIONS:
Overall Officials: Hanife Ş Ülgür, MD, Principal Investigator — University of Health Sciences, Umraniye Education and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Pendik Medipol University Hospital, Istanbul, Pendik
  - University of Health Sciences Umraniye Education and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riss S, Weiser FA, Schwameis K, Riss T, Mittlbock M, Steiner G, Stift A. The prevalence of hemorrhoids in adults. Int J Colorectal Dis. 2012 Feb;27(2):215-20. doi: 10.1007/s00384-011-1316-3. Epub 2011 Sep 20. PMID 21932016
- [Background] Maloku H, Gashi Z, Lazovic R, Islami H, Juniku-Shkololli A. Laser Hemorrhoidoplasty Procedure vs Open Surgical Hemorrhoidectomy: a Trial Comparing 2 Treatments for Hemorrhoids of Third and Fourth Degree. Acta Inform Med. 2014 Dec;22(6):365-7. doi: 10.5455/aim.2014.22.365-367. Epub 2014 Dec 19. PMID 25684841
- [Background] Pucher PH, Qurashi M, Howell AM, Faiz O, Ziprin P, Darzi A, Sodergren MH. Development and validation of a symptom-based severity score for haemorrhoidal disease: the Sodergren score. Colorectal Dis. 2015 Jul;17(7):612-8. doi: 10.1111/codi.12903. PMID 25603811
- [Background] Eddama MMR, Everson M, Renshaw S, Taj T, Boulton R, Crosbie J, Cohen CR. Radiofrequency ablation for the treatment of haemorrhoidal disease: a minimally invasive and effective treatment modality. Tech Coloproctol. 2019 Aug;23(8):769-774. doi: 10.1007/s10151-019-02054-2. Epub 2019 Aug 9. PMID 31399891
- [Background] Giamundo P, Salfi R, Geraci M, Tibaldi L, Murru L, Valente M. The hemorrhoid laser procedure technique vs rubber band ligation: a randomized trial comparing 2 mini-invasive treatments for second- and third-degree hemorrhoids. Dis Colon Rectum. 2011 Jun;54(6):693-8. doi: 10.1007/DCR.0b013e3182112d58. PMID 21552053